CLINICAL TRIAL: NCT04406857
Title: A Phase 1 Study of IPdR in Combination With Capecitabine and Radiotherapy in Rectal Cancer
Brief Title: Testing the Addition of a Radiation Sensitizing Drug, IPdR, to the Usual Chemotherapy Treatment (Capecitabine) During Radiation Therapy for Rectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03610; NCI-2020-03610 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10410 (Other: Ohio State University Comprehensive Cancer Center LAO); 10410 (Other: CTEP); UM1CA186644 (NIH); UM1CA186712 (NIH); UM1CA186716 (NIH)
Record Dates: First submitted 2020-05-28; First posted 2020-05-29 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Locally Advanced Rectal Carcinoma; Rectal Adenocarcinoma; Stage II Rectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Radiotherapy; Radiation; ropidoxuridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ropidoxuridine, capecitabine, radiation therapy) (Experimental): Patients receive ropidoxuridine PO QD over 7 days per week and capecitabine PO BID over 6 days per week for 6 weeks. Patients also undergo radiation therapy over 1 fraction per day for 5 days per week (Monday-Friday) during weeks 1-5 and for 3 days during week 6 in the absence of disease progression or unacceptable toxicity. Approximately 8-12 weeks after completion of treatment with ropidoxuridine, capecitabine, and radiation therapy, patients undergo standard of care surgery.
  Interventions: Drug: Capecitabine; Radiation: Radiation Therapy; Drug: Ropidoxuridine

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Ropidoxuridine — Given PO
  Other Names: 5-Iodo-2-pyrimidinone 2' deoxyribonucleoside; 5-Iodo-2-pyrimidinone-2'-deoxyribose; IPdR

SUMMARY:
This phase I trial studies the side effects and best dose of ropidoxuridine and how well it works when added to the usual chemotherapy treatment (capecitabine) during radiation therapy for the treatment of patients with stage II-III rectal cancer. Ropidoxuridine may help radiation therapy work better by making cancer cells more sensitive to the radiation therapy. Chemotherapy drugs, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. This study is being done to find out whether ropidoxuridine in addition to capecitabine and radiation therapy works better in treating patients with rectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of oral (PO) ropidoxuridine (IPdR) when administered with capecitabine (825 mg/m^2 twice daily [BID]) and radiation therapy (RT) (50.4 Gy in 28 fractions).

II. To determine the toxicities Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5 of the combined modality therapy, IPdR + capecitabine + RT.

SECONDARY OBJECTIVES:

I. To establish the pharmacokinetics (PK) of once daily (QD) IPdR when combined with capecitabine.

II. To evaluate iododeoxyuridine (IUdR) incorporation in circulating granulocytes and correlate these levels with IPdR plasma PK and clinical/laboratory toxicities.

III. To assess IUdR incorporation in tumor cells obtained from the surgical resection specimen and correlate IUdR incorporation in tumor cells with IPdR PK.

IV. To assess IUdR incorporation in tumor cells obtained from the surgical resection specimen and correlate IUdR incorporation in tumor cells with tumor response as measured by pathological complete response (pCR) rate and neoadjuvant rectal (NAR) score.

V. To determine the pCR rate of IPdR + capecitabine + RT at the IPdR MTD as a measure of anti-tumor activity.

VI. To determine the NAR score of IPdR + capecitabine + RT at the IPdR MTD.

EXPLORATORY OBJECTIVES:

I. To explore the relationship between extent of exposure to RT and the development and severity of adverse events.

II. To explore the drug/drug/metabolite interactions between capecitabine, IPdR, and their metabolites.

OUTLINE: This is a phase IA, dose-escalation study of ropidoxuridine followed by a phase IB study.

Patients receive ropidoxuridine PO QD over 7 days per week and capecitabine PO BID over 6 days per week for 6 weeks. Patients also undergo radiation therapy over 1 fraction per day for 5 days per week (Monday-Friday) during weeks 1-5 and for 3 days during week 6 in the absence of disease progression or unacceptable toxicity. Approximately 8-12 weeks after completion of treatment with ropidoxuridine, capecitabine, and radiation therapy, patients undergo standard of care surgery.

After completion of study treatment, patients are followed up at 4 and 8-12 weeks following chemoradiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* At diagnosis, patients must have had histologically proven adenocarcinoma of the rectum with no evidence of distant metastases
* At diagnosis, the major portion of the tumor must have been intact, and the following must be documented:

  * Distance of the lowest tumor margin from the anal verge; and
  * Intent for sphincter sparing or non-sphincter sparing surgical resection according to the primary surgeon; and
  * The majority of the untreated tumor must be < 12 cm from the anal verge or below the peritoneal reflection as determined by the treating surgeon
* At diagnosis, the tumor must have been locally advanced stage II (T3-4 N0) or stage III (N positive [+]) rectal cancer with at least one of the following:

  * Distal location (as defined by measurement on magnetic resonance imaging [MRI], endorectal ultrasound [ERUS]/pelvic computed tomography [CT] [with intravenous (IV) contrast] scan or palpable on digital rectal exam [DRE]): cT3-4 =< 5 cm from the anal verge, any N
  * Bulky: Any cT4 or evidence that the tumor is adjacent to (defined as within 3 mm of) the mesorectal fascia on MRI or ERUS/pelvic CT (with IV contrast) scan
  * High risk for metastatic disease with 4 or more regional lymph nodes (cN2). Clinical Nodal or "cN" status for eligibility includes the total number of nodes (N2 = 4 or more) in the mesorectal and superior rectal stations measuring >= 1.0 cm in any axis on cross sectional or endoscopic imaging. Nodes must measure 1.0 cm or greater to be considered positive for this eligibility requirement
  * Not a candidate for sphincter-sparing surgical resection prior to neoadjuvant therapy (as planned by the primary surgeon)
* Patients must have received 8 cycles of neoadjuvant leucovorin, fluorouracil, and oxaliplatin (mFOLFOX) and must have completed this therapy at least 3 weeks (and no more than 6 weeks) prior to enrollment on this study
* Patients must intend to undergo surgical resection of the rectal primary tumor following chemoradiotherapy
* Age >= 18 years

  * Because no dosing or adverse event (AE) data are currently available on the use of IPdR in combination with capecitabine and RT in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,200/mcL
* Platelets >= 100,000/mcL
* Hemoglobin > 10 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x institutional ULN
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Creatinine =< 1.5 x institutional ULN OR glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2
* Alkaline phosphatase =< 3 x institutional ULN
* Sodium, potassium, chloride, bicarbonate, and magnesium within institutional normal limits
* Patients with acquired immunodeficiency syndrome (acquired immunodeficiency syndrome [AIDS]-related illnesses) or known human immunodeficiency virus (HIV) disease must:

  * Have a CD4 count >= 200 cells/uL within 30 days before enrollment,
  * Be off all antiretroviral therapy (prophylaxis/treatment) more than 60 days before enrollment, and
  * Have no evidence of opportunistic infections
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured and be receiving no therapy
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this trial, patients should be class 2B or better
* Patients must have the ability to swallow and retain oral medication
* The effects of IPdR on the developing human fetus are unknown. For this reason and because radiosensitizing agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential (WOCBP)* and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. WOCBP must have a negative urine or serum pregnancy test within 72 hours prior to enrollment. If urine pregnancy results are positive or cannot be confirmed as negative, a serum pregnancy test will be required. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of IPdR administration

  * Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior mFOLFOX6 chemotherapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* Patients with impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral IPdR and capecitabine (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). Patients with active inflammatory bowel disease (i.e., patients requiring current medical interventions or who are symptomatic) or have a history of abdominal surgery or other medical condition that may, in the opinion of the treating physician, interfere with GI motility or absorption. Patients with colostomies are allowed unless colostomy is for one of the precluded reasons above
* Treatment with warfarin is not allowed. However, therapy with heparin, low molecular weight heparin (LMWH), and DOACs (direct oral anticoagulating agent) such as dabigatran (Pradaxa), rivaroxaban, and apixaban (Eliquis) is allowed
* Patients with an active concurrent invasive malignancy
* History of prior invasive rectal malignancy, regardless of disease-free interval
* Patients who have received pelvic RT for rectal cancer, or prior pelvic RT for any other malignancy that would prevent the patient from receiving the required RT for this study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to IPdR or capecitabine
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because IPdR may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with IPdR, breastfeeding should be discontinued if the mother is treated with IPdR. These potential risks may also apply to other agents used in this study
* Patients that received live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal flu vaccines that do not contain live virus are permitted
* Known homozygous DPD (dihydro pyrimidine dehydrogenase) deficiency
* History of, or any evidence of, active non-infectious pneumonitis
* Active autoimmune disease that has required systemic treatment within the past 2 years (i.e., with use of modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* History of active TB (Bacillus tuberculosis)
* Active or chronic infection requiring systemic therapy
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study therapy. The use of physiologic doses of corticosteroids may be approved after consultation with the study principal investigator (PI)
* Active seizure disorder uncontrolled by medication
* Synchronous colon cancer
* Other invasive malignancy within 5 years. Exceptions are colonic polyps, non-melanoma skin cancer, or carcinoma-in-situ of the cervix
* Antineoplastic therapy (e.g., chemotherapy or targeted therapy) for other invasive malignancy within 5 years (for the purposes of this study hormonal therapy is not considered chemotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kunos, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (9):
- United States (9):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Kunos CA, Piekarz R, Collins JM, Kinsella TJ. A case report of typhlitis during novel use of ropidoxuridine-capecitabine-radiotherapy for treatment-naive rectal cancer. Cancer Chemother Pharmacol. 2023 Aug;92(2):151-155. doi: 10.1007/s00280-023-04561-4. Epub 2023 Jun 27. PMID 37369852

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose
Description: The maximum-tolerated dose is defined as the dose below which 2 or more of 6 patients experience dose-limiting toxicities attributable to ropidoxuridine.
Time Frame: Up to 38 days
Population: Data not collect and analyzed
Arm/Group | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy)
Number analyzed (Participants) | 0

2. Primary Outcome: Incidence of Dose-limiting Toxicities (Part IB)
Description: Assessed by Common Terminology Criteria for Adverse Events version 5 and reached when any two grade 3 treatment-related non-hematologic toxicities or one grade 4 treatment-related hematologic and/or gastrointestinal toxicity are observed in two of the 6 patients enrolled at that dose level.
Time Frame: Up to 38 days
Population: Data not collect and analyzed
Arm/Group | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Tissue Biomarker Levels
Description: Will be measured on continuous and binary scales will be assessed using Wilcoxon signed rank or McNemar's tests, respectively (two-sided; alpha = 0.05). Associations between therapeutic response and baseline biomarker values or temporal changes in biomarkers will be explored using Fisher's exact tests or Wilcoxon rank sum tests.
Time Frame: Baseline up to 8-12 weeks following completion of chemotherapy
Population: Data not collect and analyzed
Arm/Group | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Ropidoxuridine Incorporation in Circulating Granulocytes
Description: Will correlate these levels with ropidoxuridine plasma pharmacokinetics. Two-sided Fisher's z-test with significance level of 0.05 and power of 80% will be used and the study will reject the null hypothesis (lack of correlation or r0 = 0) if we observe a correlation with r ranging from 0.79 for N = 10 subjects to 0.49 for N = 30 subjects.
Time Frame: Prior to ropidoxuridine dose and at 30, 60, 120, and 240 minutes after ropidoxuridine dose on day 8, then at 1-2 hours after ropidoxuridine dose on days 21 and 35
Population: Data not collect and analyzed
Arm/Group | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Percentage of Ropidoxuridine Incorporation in Circulating Granulocytes, Peripheral Blood Counts, and Toxicities
Description: For the correlation of percentage of ropidoxuridine deoxyribonucleic acid incorporation in circulating granulocytes and peripheral blood counts and toxicities, assuming the target prevalence of grade 3/4 toxicity of 30%, the study will have a power of 80% with significance level of 0.05 on a two-sample means test to rule out the null hypothesis (equal means in groups with/ without grade 3/4 toxicity, m0 = m1) if the observed mean percentage of ropidoxuridine-deoxyribonucleic acid incorporation for patients with grade 3/4 toxicity is m1 = 3.3 times the mean m0 in the other group for N = 10 enrolled subjects, and m1 = 2.1 times the mean m0 for N = 30.
Time Frame: Prior to the ropidoxuridine on day 8, and at 1-2 hours following the ropidoxuridine dose on days 21 and 35
Population: Data not collect and analyzed
Arm/Group | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: Pathological Complete Response Rate at the Maximum-tolerated Dose
Description: In rectal cancer, the absence of viable tumor cells in the resection specimen (primary tumor mass, surrounding tissue and lymph nodes, T0 N0 M0) at the time of surgery, termed pathologic complete response. Pathologic complete response determination will be made by the pathologist at the treating institution.
Time Frame: At the time of surgery
Population: Data not collect and analyzed
Arm/Group | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Neoadjuvant Rectal Score at the Maximum-tolerated Dose
Description: Neoadjuvant rectal score is calculated based on the clinical T stage (cT), pathological T (pT) and pN stages as neoadjuvant rectal score = [5pN- 3 (cT- pT) + 12]2 / 9.61.
Time Frame: At 6-10 weeks following completion of therapy
Population: Data not collect and analyzed
Arm/Group | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Relationship Between Extent of Exposure to Radiotherapy and Incidence and Severity of Adverse Events
Time Frame: Up to 3 years
Population: Data not collect and analyzed
Arm/Group | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Interactions of Capecitabine, IPdR and Their Metabolites
Time Frame: Up to 3 years
Population: Data not collect and analyzed
Arm/Group | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected and graded from baseline until completion of the study up to 1 year.
Arm/Group | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ropidoxuridine, Capecitabine, Radiation Therapy) (N=1)
Cecal inflammation (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial had inadequate accrual rate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT04406857/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT04406857/ICF_001.pdf